CLINICAL TRIAL: NCT03551119
Title: Physical Activity in Renal Disease (PAIRED): A Randomized Controlled Trial of the Effect on Hypertension
Brief Title: Physical Activity in Renal Disease (PAIRED): The Effect on Hypertension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Stephanie Thompson, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00078564
Record Dates: First submitted 2018-05-12; First posted 2018-06-11 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: In this parallel arm control trial, participants recruited from outpatient CKD clinics in Alberta Kidney Care North, Edmonton, Alberta, Canada will be randomized (1:1) to enhanced usual care (measurement of physical activity levels) or an exercise intervention.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants cannot be blinded to group assignment; however, the primary outcome is objectively measured (24-hour ambulatory blood pressure measurement). For main trial secondary outcomes, assessors will be blinded to allocation status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Personnel experienced in training people with chronic conditions (exercise specialist) will supervise the exercise training. At each in-center session in phase 1, the patient's exercise will be monitored to assess whether they are achieving target levels. Training intensities will be prescribed based on the most recent exercise test.
  Phase 1: an eight-week program of once weekly-supervised facility-based exercise sessions and twice weekly home-based sessions.
  Phase 2: a 16-week home-based exercise program overseen by an exercise specialist. During this phase, participants will be progressed through their home-based exercise program from Phase 1 on an individual basis.
  i. Frequency. A minimum of three exercise sessions per week. ii. Intensity. A moderate intensity (40-60% heart rate reserve) based on exercise testing.
  iii. Time. 150 minutes of exercise per week. iv. Type. We will prescribe aerobic exercise supplemented with isometric resistance exercises.
  Interventions: Behavioral: Exercise
- Enhanced usual care (Other): Participants in the control group will perform accelerometry. This is enhanced usual care because physical activity measurement is not routinely performed in CKD clinics. Control arm participants will only receive their accelerometry data after they have completed the study.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: Exercise — See previous description
  Arms: Exercise
Other: Enhanced usual care — See previous description
  Arms: Enhanced usual care

SUMMARY:
Background and importance: Hypertension is highly prevalent among Canadians with non-dialysis dependent chronic kidney disease (CKD). It is a modifiable risk factor for both cardiovascular (CV) events and CKD progression. Exercise is an effective strategy for blood pressure (BP) reduction in the general population but in people with CKD, hypertension is mediated by different causes (i.e. vascular stiffness, volume expansion) and it is unclear whether exercise will reduce BP in this population. Consequently, exercise resources are not offered in the routine multidisciplinary care of people with CKD and the prevalence of sedentary behaviour remains double that of the general population. The role of exercise in CKD management is also an important question for patients. From CIHR-supported workshops with patients, the role of lifestyle, such as exercise in CKD was a top research priority.

Research aims: i.To determine the effect of exercise on mean ambulatory systolic blood pressure (SBP) in people with CKD compared to usual care. The investigators hypothesize that exercise training will significantly reduce BP compared to control. ii.To inform the design of a larger, multi-center trial evaluating the effect of exercise on the risk of CKD progression.

Methods: A 160 participant, single center randomized trial of adults from Alberta Kidney Care North CKD clinics, Edmonton, Albert, Canada. Participants with an estimated glomerular filtration rate (eGFR) of 15-44 ml/min per 1.73m2 and SBP >130 mmHg will be randomized, stratified by eGFR (<30 versus ≥ 30) to an exercise intervention or usual care. The main outcome is the difference in 24-hour ambulatory SBP after eight weeks of exercise training between groups. Secondary outcomes include: BPs at eight and 24 weeks, dose of anti-hypertensives, aortic stiffness, CV-risk markers, CV fitness, 7-day accelerometry, quality of life, safety, and in an exploratory analysis, eGFR and proteinuria. The intervention is thrice weekly moderate intensity aerobic exercise supplemented with isometric resistance exercise, targeting 150 minutes per week and delivered over 24-weeks. Phase 1: one supervised weekly sessions and home-based sessions (eight weeks). Phase 2: home-based sessions (16 weeks). To detect a clinically important BP reduction of 5 mmHg between groups requires 128 patients (two sample t-test, alpha 0.05, beta 0.2, common standard deviation of 10 mmHg). Assuming 20% dropout requires 160 patients. For the primary outcome, the investigators will use a mixed linear regression model in which BP is regressed on group, baseline SBP and eGFR, and time point.

Expected outcomes: The findings from this study will address a significant knowledge gap in hypertension management in CKD, inform care-delivery and the design of a larger study on CKD progression. This proposal aligns with priorities for both patients and decision makers: to identify the role of exercise in CKD management and to reshape the delivery of renal care so that it is more consistent with patient values and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Resting SBP >120 mmHg systolic on screening BP clinic measurements (with an electronic sphygmomanometer, mean of three readings after first reading is discarded) and at least one previous SBP measurement above 120 mmHg on a separate occasion within the past six months (home or clinic measurement).
* Stable on blood pressure medications for the past eight weeks
* eGFR 15-44 ml/min per 1.73m2 eGFR between 15-44 ml/min per 1.73m2 within the last three months and one additional value in this rage in the last 12 months.
* Independent ambulation with or without an assistive device for at least three consecutive minutes
* Cognition and English language sufficient enough to understand written information, provide consent, and comply with the testing and interventions
* Approval of the attending nephrologist
* No significant exercise-induced arrhythmia or new ischemia on submaximal incremental exercise testing (final screening step)

Exclusion Criteria:

* Resting SBP >160 mmHg or DBP > 110 mmHg on screening BP clinic measurement (Note: the individual may be re-screened 8 weeks after medication adjustment)
* Arm circumference greater than 54 centimeters (size limit of large ABPM cuff)
* Recent (<6 weeks) or planned (<6 months) major cardiovascular events or procedures
* Any known contraindication to exercise (American College of Sports Medicine Guidelines)

Acute myocardial infarction (3-5 days) or unstable angina; Uncontrolled symptomatic arrhythmias; Active endocarditis; Acute myocarditis or pericarditis; Symptomatic severe aortic stenosis; Acute pulmonary embolism or deep vein thrombosis; Suspected dissecting aneurysm; Uncontrolled asthma; Uncontrolled pulmonary edema; Room air desaturation to <85%; Acute non-cardiopulmonary disorder that may affect exercise performance (infection, orthopedic problem); Mental impairment leading to inability to cooperate; Uncontrolled hypertension (as above)

* Pregnant or planning to become pregnant
* Transplant
* Life expectancy or predicted time to renal replacement therapy <9 months (attending physician judgment)
* Planned move or hospital admission within the next 9 months
* Currently enrolled in an interventional clinical trial; currently enrolled in a structured exercise program or performing regular exercise training > 2 day/week in the last 3 months
* Taking other medications known to affect blood pressure (prednisone cyclosporine) and expected adjustment in the next 9 months
* Significant barrier to participation in a home exercise program or an insurmountable barrier to attend in-center training sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory SBP | 8 weeks
  mean 24-hour ambulatory systolic blood pressure

SECONDARY OUTCOMES:
antihypertensive use | 8 and 24 weeks
  Using the assigned DDD (WHO) for that drug
KDQOL-36 | 8 and 24 weeks
  Kidney Disease and Quality of Life instrument - this is a short form that includes the SF-12 plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF
IPAQ-SF | 8 and 24 weeks
  International Physical Activity Questionnaire - Short Form
SEE scale | 8 and 24 weeks
  Self Efficacy for Exercise questionnaire - the total score ranges from 0 to 90. High scores indicate higher self-efficacy in exercise. There are 9 questions; responses vary from 0 to 10. The mean score on each question is 5.5.
EQ-5D | 8 and 24 weeks
  European Quality of Life (EuroQOL) health questionnaire with 5 dimensions
pulse wave velocity | 8 and 24 weeks
  measurement of aortic stiffness (femoral carotid, radial carotid)
body mass index | 8 and 24 weeks
  calculated as weight in kilograms divided by height in meters squared
Fat mass | 8 and 24 weeks
  Body composition using bioimpedance spectroscopy
clinic blood pressure | 8 and 24 weeks
  with a oscillometric sphygmomanometer
Oxygen uptake (VO2 peak) | 8 and 24 weeks
  Cardiopulmonary exercise testing
estimated glomerular filtration rate | 8 and 24 weeks
c-reactive protein | 8 and 24 weeks
total cholesterol | 8 and 24 weeks
LDL | 8 and 24 weeks
HDL | 8 and 24 weeks
triglycerides | 8 and 24 weeks
HgA1C | 24 weeks
  glycated hemoglobin
spot urinary sodium | 8 and 24 weeks
  measured on a non-exercise day
spot urinary protein | 8 and 24 weeks
  measured on a non-exercise day
7-day accelerometry | 8 and 24 weeks
  number of steps
7-day accelerometry | 8 and 24 weeks
  sedentary time
7-day accelerometry | 8 and 24 weeks
  time in light activity
7-day accelerometry | 8 and 24 weeks
  time in moderate activity
7-day accelerometry | 8 and 24 weeks
  time in vigorous activity
7-day accelerometry | 8 and 24 weeks
  time in very vigorous activity
7-day accelerometry | 8 and 24 weeks
  METS
7-day accelerometry | 8 and 24 weeks
  sedentary bouts
24-hour ABPM | 8 and 24 weeks
  daytime, night time systolic and diastolic BP
Adherence | 8 and 24 weeks
  70% of in centre sessions attended and 70% of home sessions performed prescribed (accelerometry and log book)
Body cell mass | 8 and 24 weeks
  Body composition using bioimpedance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Thompson, MD PhD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, outpatient dialysis unit, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta

REFERENCES:
- [Derived] Thompson S, Wiebe N, Gyenes G, Davies R, Radhakrishnan J, Graham M. Physical Activity In Renal Disease (PAIRED) and the effect on hypertension: study protocol for a randomized controlled trial. Trials. 2019 Feb 8;20(1):109. doi: 10.1186/s13063-019-3235-5. PMID 30736832